CLINICAL TRIAL: NCT05624450
Title: A Phase III, Multicentre, Randomised, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Tozorakimab (MEDI3506) in Patients Hospitalised for Viral Lung Infection Requiring Supplemental Oxygen
Brief Title: Efficacy and Safety of Tozorakimab in Patients Hospitalised for Viral Lung Infection Requiring Supplemental Oxygen
Acronym: TILIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9185C00001; 2023-507031-38-00 (Registry Identifier: CTIS); 2022-003107-15 (EudraCT Number)
Record Dates: First submitted 2022-11-11; First posted 2022-11-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Viral Lung Infection and Acute Respiratory Failure
Keywords: Acute Respiratory Failure; Acute Respiratory Distress Syndrome; Viral lung infection; Tozorakimab; Supplemental Oxygen; IL-33; COVID-19; SARS-CoV-2; Coronavirus Infections; Virus Diseases; SARS Coronavirus; MEDI3506; Respiratory Tract Infections; Infections; Lung Diseases; Influenza
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19; Coronavirus Infections; Virus Diseases; Severe Acute Respiratory Syndrome; Respiratory Tract Infections; Infections; Lung Diseases; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tozorakimab (Experimental): Approximately 2870 participants will be randomized in a 1:1 ratio. Arm 1 (n=approximately 1435) will receive a single dose of tozorakimab.
  Interventions: Drug: Tozorakimab
- Placebo (Placebo Comparator): Approximately 2870 participants will be randomized in a 1:1 ratio. Arm 2 (n=approximately 1435) will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tozorakimab — Single IV dose of tozorakimab on Day 1.
  Other Names: MEDI3506
  Arms: Tozorakimab
Drug: Placebo — Single IV dose of matching placebo on Day 1.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of tozorakimab, as an add-on to SoC in patients with viral lung infection requiring supplemental oxygen, on the prevention of death or progression to IMV/ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥ 18 years old at the time of signing the informed consent form.
* Patients hospitalised with viral lung infection.
* Hypoxaemia requiring treatment with supplemental O2.

Hypoxaemia is defined as:

SpO2 ≤ 90% OR

SpO2 ≤ 92% AND one or both of the following:

Radiographic infiltrates by CXR/CT compatible with viral lung infection per investigator judgement.

Use of accessory muscles of respiration or RR (respiratory rate) > 22.

- Patient remains hypoxaemic at randomisation requiring treatment with supplemental oxygen.

Exclusion Criteria:

* Known fungal or parasitic lung infection, aspiration lung infection, lung abscess, or evidence of septic shock. Bacterial co-infection is allowed, unless, in the opinion of the investigator, bacterial infection defines the severity of the participant's condition.
* Hypoxaemia caused primarily by extrapulmonary insult or by lung injury of non-infective aetiology.
* Ongoing IMV/ECMO at randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2870 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who die or progress to Invasive Mechanical Ventilation (IMV) / Extracorporeal Membrane Oxygen (ECMO) | by Day 28
  To evaluate the effect of tozorakimab versus placebo as an add on to Standard of Care (SoC) in participants with viral lung infection requiring supplemental oxygen on the prevention of death or progression to IMV/ECMO.

SECONDARY OUTCOMES:
Proportion of participants who die | by Day 60
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on all-cause mortality.
Number of days alive and outside of Intensive Care Unit (ICU) | over 28 day period
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on ICU stay.
Number of days alive and free of supplemental oxygen | over 28 day period
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on the duration of oxygen supplementation.
Time to death or progression to Invasive Mechanical Ventilation (IMV) / Extracorporeal Membrane Oxygen (ECMO) | over 28 day and 60 day period
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on prolonging time to death or IMV/ECMO.
Proportion of participants who die or progress to Invasive Mechanical Ventilation (IMV) / Extracorporeal Membrane Oxygen (ECMO) | by Day 60
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on prolonging time to death or IMV/ECMO.
Time to death (all cause) | over 28 day and 60 day period
  To evaluate the effect of Tozorakimab versus Placebo as add-on to Standard of Care (SoC) on prolonging time to death.
Proportion of participants who die | by Day 28
  To evaluate the effect of Tozorakimab versus Placebo as add-on to Standard of Care (SoC) on prolonging time to death.
Number of days alive and free of Invasive Mechanical Ventilation (IMV) / Extracorporeal Membrane Oxygen (ECMO) | over 28 day and 60 day period
  To evaluate the effect of Tozorakimab versus placebo as add-on to Standard of Care (SoC) on ventilator use.
Number of days alive and ventilator free | over 28 day and 60 day period
  To evaluate the effect of Tozorakimab versus placebo as add-on to Standard of Care (SoC) on ventilator use.
Proportion of participants with Intensive Care Unit (ICU) admission or death | by Day 28
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on ICU admissions.
Proportion of participants with Intensive Care Unit (ICU) admission or death | by Day 60
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on ICU admissions.
Proportion of participants alive and discharged | by Day 28
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on duration of hospitalisation.
Proportion of participants alive and discharged | by Day 60
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on duration of hospitalisation.
Time to discharge | over 28 day and 60 day period
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on duration of hospitalisation.
Time to being off supplemental oxygen | over 28 day and 60 day period
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on duration of hospitalisation.
World Health Organization (WHO) 10-category ordinal Clinical Progression Scale | by Day 60
  To evaluate the effect of tozorakimab versus placebo as add-on to Standard of Care (SoC) on clinical status as assessed by the Investigator using WHO 10-category ordinal Clinical Progression Scale (0 least severe to 10 most severe).
Presence of anti-drug antibodies | over 60 day period
  To evaluate the immunogenicity (presence of tozorakimab anti-drug antibodies in blood serum) in participants with viral lung infection requiring supplemental oxygen.
Baseline serum interleukin-33/soluble Suppression of Tumorgenicity 2 (IL-33/sST2) complex levels relative to primary endpoint | Day 1
  To evaluate the use of baseline serum IL-33/sST2 complex levels (U/mL) to predict treatment response with tozorakimab versus placebo as add on to Standard of Care (SoC).

CONTACTS AND LOCATIONS:
Locations (363):
- United States (63):
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Chula Vista, California
  - Research Site, Fresno, California
  - Research Site, La Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Torrance, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Bradenton, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, South Pasadena, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Elmhurst, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, Springfield, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Saint Paul, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Potsdam, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Corvallis, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Greenville, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Green Bay, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (6):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Munro
  - Research Site, Rosario
- Australia (5):
  - Research Site, Adelaide
  - Research Site, Bedford Park
  - Research Site, New Lambton Heights
  - Research Site, Port Macquarie
  - Research Site, South Brisbane
- Belgium (4):
  - Research Site, Kortrijk
  - Research Site, Ottignies
  - Research Site, Roeselare
  - Research Site, Yvoir
- Brazil (17):
  - Research Site, Belo Horizonte
  - Research Site, Campinas
  - Research Site, Caxias do Sul
  - Research Site, Curitiba
  - Research Site, Indaiatuba
  - Research Site, Jaú
  - Research Site, Natal
  - Research Site, Niterói
  - Research Site, Passo Fundo
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Caetano do Sul
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (6):
  - Research Site, Montana
  - Research Site, Pernik
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Canada (10):
  - Research Site, Calgary, Alberta
  - Research Site, New Westminster, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Brampton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
- China (22):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuyang
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jining
  - Research Site, Nanchang
  - Research Site, Nantong
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Weifang
  - Research Site, Wuhan
  - Research Site, Yantai
  - Research Site, Yinchuan
  - Research Site, Yueyang
  - Research Site, Zhengzhou
- Colombia (5):
  - Research Site, Bogota DC
  - Research Site, Floridablanca
  - Research Site, Medellín
  - Research Site, Soledad
  - Research Site, Villavicencio
- Czechia (7):
  - Research Site, Benešov
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Kolín
  - Research Site, Kyjov
  - Research Site, Mladá Boleslav
  - Research Site, Prague
- Denmark (10):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Copenhagen
  - Research Site, Copenhagen Ø
  - Research Site, Herning
  - Research Site, Hillerød
  - Research Site, Hvidovre
  - Research Site, Kolding
  - Research Site, Odense C
  - Research Site, Vejle
- Egypt (3):
  - Research Site, Alexandria
  - Research Site, Cairo
  - Research Site, New Cairo
- France (12):
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, La Tronche
  - Research Site, Le Coudray
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Orléans
  - Research Site, Strasbourg
  - Research Site, Tours
- Germany (11):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Kiel
  - Research Site, Leverkusen
  - Research Site, Marburg
  - Research Site, Regensburg
  - Research Site, Rosenheim
  - Research Site, Rostock
- Greece (5):
  - Research Site, Athens
  - Research Site, Exohi Thessaloniki
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Hungary (7):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kistarcsa
  - Research Site, Nyíregyháza
  - Research Site, Pécs
- India (12):
  - Research Site, Ahmedabad
  - Research Site, Belagavi
  - Research Site, Chennai
  - Research Site, Gurugram
  - Research Site, Gūrgaon
  - Research Site, Hyderabad
  - Research Site, Kanpur
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Thane
  - Research Site, Vijayawada
- Israel (9):
  - Research Site, Afula
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
- Italy (6):
  - Research Site, Arezzo
  - Research Site, Brescia
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Torino
- Japan (38):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Gifu
  - Research Site, Ginowan-shi
  - Research Site, Hanyu-shi
  - Research Site, Hiroshima
  - Research Site, Hitachi-shi
  - Research Site, Isehara-shi
  - Research Site, Izumisano
  - Research Site, Izumo-shi
  - Research Site, Kamakura-shi
  - Research Site, Kamogawa-shi
  - Research Site, Kanazawa
  - Research Site, Kasuga-shi
  - Research Site, Kawasaki-shi
  - Research Site, Koshigaya-shi
  - Research Site, Kumagaya-shi
  - Research Site, Kumamoto
  - Research Site, Kusatsu-shi
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Meguro-ku
  - Research Site, Mitaka-shi
  - Research Site, Nagoya
  - Research Site, Nerima-ku
  - Research Site, Okayama
  - Research Site, Okazaki-shi
  - Research Site, Omuta-shi
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Tachikawa-shi
  - Research Site, Takamatsu
  - Research Site, Urasoe-shi
  - Research Site, Ureshino-shi
  - Research Site, Yokohama
- Malaysia (11):
  - Research Site, Kota Kinabalu
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Terengganu
  - Research Site, Kuantan
  - Research Site, Kubang Kerian
  - Research Site, Malacca
  - Research Site, Petaling Jaya
  - Research Site, Pulau Pinang
  - Research Site, Sarawak Miri
  - Research Site, Selangor Darul Ehsan
  - Research Site, Shah Alam
- Mexico (7):
  - Research Site, Aguascalientes
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Monterrey
  - Research Site, San Luis Potosí City
  - Research Site, Tlalpan
  - Research Site, Xalapa
- Peru (4):
  - Research Site, Cusco
  - Research Site, El Agustino
  - Research Site, Lima
  - Research Site, Piura
- Philippines (4):
  - Research Site, Cebu
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (7):
  - Research Site, Chrzanów
  - Research Site, Lodz
  - Research Site, Rzeszów
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Łańcut
  - Research Site, Łęczna
- Research Site, Bayamón, Puerto Rico
- Romania (6):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Iași
  - Research Site, Sibiu
  - Research Site, Timișoara
- Saudi Arabia (2):
  - Research Site, Jeddah
  - Research Site, Riyadh
- Research Site, Bratislava, Slovakia
- South Africa (4):
  - Research Site, Johannesburg, Soweto
  - Research Site, Observatory
  - Research Site, Parktown
  - Research Site, Westdene
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Jeonju
  - Research Site, Seoul
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Ourense
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Santander
  - Research Site, Valencia
- Sweden (8):
  - Research Site, Helsingborg
  - Research Site, Huddinge
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Solna
  - Research Site, Stockholm
  - Research Site, Umeå
  - Research Site, Västerås
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan
  - Research Site, Taoyuan District
- Thailand (7):
  - Research Site, Bangkok
  - Research Site, Banphaeo
  - Research Site, Chiang Mai
  - Research Site, Khlong Luang
  - Research Site, Khon Kaen
  - Research Site, Phutthamonthon
  - Research Site, Ubonratchathani
- Turkey (Türkiye) (7):
  - Research Site, Ankara
  - Research Site, Diyarbakır
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, İzmit
  - Research Site, Malatya
  - Research Site, Ortahisar
- United Kingdom (12):
  - Research Site, Bristol
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Hampshire
  - Research Site, Huddersfield
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Oxford
  - Research Site, Prescot
  - Research Site, Tyne and Wear
  - Research Site, Wythenshawe
- Vietnam (5):
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh City
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home